CLINICAL TRIAL: NCT07009795
Title: Rise & Renew (Remembering, Expressing, Navigating, Embracing, Witnessing): Enhancing Well-being Among Black Women Who've Experienced a First-order Bereavement Event
Brief Title: Rise & Renew: Supporting Well-Being in Black Women After the Loss of a Loved One
Acronym: RENEW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lillian Haley, PhD (Industry)
Collaborators: The Good Stewards Partnership (Unknown)
Responsible Party: Sponsor-Investigator, Lillian Haley, PhD, Principal Investigator, Haley Evaluation & Research Services
Organization: Haley Evaluation & Research Services (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RN052025
Record Dates: First submitted 2025-05-20; First posted 2025-06-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bereavement; Grief; Psychological Distress; Well Being
Keywords: Bereavement; Faith-Based Support; Community-Based Intervention; Wellness; African American Women; Spirituality; Psychosocial Support Systems; Mental Health Intervention; Holistic Healing
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two different groups:
  * Immediate Virtual Group Support: Starts the 10-week virtual program within 10 days of completing the retreat.
  * Delayed Virtual Group Support: Delays the start of the 10-week virtual program by 10 weeks.
  These two groups run in parallel, with both participating in the wellness retreat weekend, followed by different timelines for receiving the 10-week virtual support group part of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Virtual Group Support (Experimental): Receives the in-person wellness retreat and begins the 10-week virtual support phase the following weekend.
  Interventions: Behavioral: Rise & Renew Hybrid Grief Support Program
- Delayed Virtual Group Support (No Intervention): Attends the same in-person wellness retreat but does not begin the 10-week virtual support program until after a 10-week delay.

INTERVENTIONS:
Behavioral: Rise & Renew Hybrid Grief Support Program — The Rise & Renew Hybrid Grief Support Program is a culturally responsive, multi-component behavioral intervention designed specifically for Black women aged 40 and older who have experienced the loss of a spouse, parent, or child. It integrates wellness practices, grief support, spiritual care, and community healing in a hybrid format that includes both an in-person and virtual component.
  This intervention is distinguished by its cultural tailoring for middle-aged and older Black women, co-facilitation by both a trained facilitator and a faith-based leader, and its combination of expressive arts, spiritual guidance, and practical wellness strategies delivered in a hybrid format. It addresses grief holistically through emotional, physical, spiritual, and social dimensions, and emphasizes culturally relevant healing practices often overlooked in conventional grief programs.
  Arms: Immediate Virtual Group Support

SUMMARY:
This study is testing a new grief support program called Rise & Renew (Remembering, Expressing, Navigating, Embracing, Witnessing) designed for Black women ages 40 and older who have experienced the loss of a close loved one, such as a spouse or significant other, parent, or child (including pregnancies). The program includes a weekend wellness retreat followed by 10 weeks of online group support. Participants will be randomly assigned to start weekly virtual sessions right away or after a 10-week delay. The study will help the investigators learn whether the program is helpful, easy to take part in, and meaningful for those who attend. The investigators believe that a culturally tailored program that focuses on healing, wellness, and community will improve emotional health, spiritual well-being, and resilience during the grief process.

DETAILED DESCRIPTION:
Rise & Renew (Remembering, Expressing, Navigating, Embracing, Witnessing) is a pilot randomized controlled trial (RCT) using a waitlist control design to evaluate the feasibility, acceptability, and preliminary outcomes of a culturally responsive hybrid grief support program for Black women aged 40 and older who have experienced the death of a spouse/significant other, parent, or child (including pregnancies).

This study addresses critical gaps in bereavement support for Black women, who often face intersecting emotional, cultural, and spiritual needs. The Rise & Renew program is rooted in wellness practices, spiritual care, and culturally grounded healing rituals.

Study Design

After completing the baseline assessment, participants will be randomly assigned (1:1) to one of two groups using a computer-generated randomization sequence:

* Group A (Intervention Group): Will participate in an in-person weekend retreat and begin the 12-week Rise & Renew virtual support program immediately.
* Group B (Waitlist Control Group): Will attend the same in-person retreat but will delay participation in the 12-week virtual program for 12 weeks.

This staggered model allows researchers to examine short-term changes in well-being and grief outcomes while providing all participants access to the full intervention.

Intervention Description

Rise & Renew is a 12-week hybrid grief support program designed to affirm the cultural identity, spirituality, and healing traditions of Black women. The program consists of:

* One In-Person Weekend Retreat: Focused on wellness, healing rituals, community building, and expressive arts.
* 10 Weekly Virtual Support Sessions: Co-facilitated by a professional with group facilitation expertise and a Black faith leader. Session themes include:
* Grief and emotional healing
* Spiritual and personal growth
* Financial empowerment
* Self-care and wellness
* Building social support networks

Recruitment and Eligibility The study is open to self-identified Black women aged 40 and older, living in the U.S. South Region, including Alabama, Arkansas, Delaware, District of Columbia, Florida, Georgia, Kentucky, Louisiana, Maryland, Mississippi, North Carolina, Oklahoma, South Carolina, Tennessee, Texas, Virginia, and West Virginia. Recruitment will be conducted via digital outreach, including phone calls, text messages, and a study webpage.

Data Collection

This study uses a mixed-methods approach to collect both quantitative and qualitative data:

* Needs Assessment Survey: Conducted before the retreat to gather information on participants' unique needs and expectations, allowing facilitators to tailor the program accordingly.
* Baseline: Participants will complete a pre-intervention survey in Qualtrics assessing grief, stress, depression, physical wellness (including self-reported blood pressure and weight), social support, and financial resilience.
* Post-Intervention: Surveys and optional focus groups/interviews will assess perceived benefits, changes in well-being, and overall program satisfaction.

All participants will be invited to join Part 2 (10-week support group) after the retreat, regardless of initial group assignment. Participation is voluntary, and no compensation will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a Black or African American woman
* Aged 40 years or older at the time of enrollment
* Has experienced the death of a spouse, parent, or child (first-order bereavement)
* Resides in the U.S. South Region, including: Alabama, Arkansas, Delaware, District of Columbia, Florida, Georgia, Kentucky, Louisiana, Maryland, Mississippi, North Carolina, Oklahoma, South Carolina, Tennessee, Texas, Virginia, or West Virginia
* Has access to a reliable internet connection and a device capable of running Zoom
* Is able to attend a 2-day in-person retreat in the Stone Mountain, GA area
* Is able and willing to participate in 10 weekly virtual group sessions
* Provides informed consent to participate in the study
* Agrees to complete pre- and post-intervention surveys

Exclusion Criteria:

* Has not experienced the death of a spouse, parent, or child
* Under the age of 40 at the time of enrollment
* Does not reside in the U.S. South Region
* Unable to attend the in-person retreat in Stone Mountain, GA
* Unwilling or unable to participate in weekly Zoom sessions
* Does not have access to the necessary technology for virtual sessions
* Does not provide informed consent
* Currently receiving intensive psychotherapy or psychiatric treatment that would conflict with participation
* Any condition or circumstance that, in the opinion of the investigators, may compromise the participant's ability to safely engage in the group setting

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | From baseline to the end of the 10-week support group intervention
  The 4-item Feasibility of Intervention Measure was developed for evaluating the success of feasibility, demonstrating encouraging psychometric properties. The items that are scored on a scale of 0 to 4, where 0 indicates "completely disagree," and 4 indicates "completely agree". Thus, the range for each scale extends from 0 - 16, with higher scores indicating higher feasibility.
Acceptability of Intervention Measure (AIM) | FroFrom baseline to the end of the 10-week support group intervention
  The 4-item Acceptability of Intervention Measure was developed for evaluating the success of acceptability, demonstrating encouraging psychometric properties. The items are scored on a scale of 0 to 4, where 0 indicates "completely disagree," and 4 indicates "completely agree". Thus, the range for each scale extends from 0 - 16, with higher scores indicating higher acceptability.
Intervention Appropriateness Measure (IAM) | From baseline to the end of the 10-week support group intervention
  The 4-item Acceptability of Intervention Measure was developed for measuring the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. The items are scored on a scale of 0 to 4, where 0 indicates "completely disagree," and 4 indicates "completely agree". Thus, the range for each scale extends from 0 - 16, with higher scores indicating higher appropriateness.

SECONDARY OUTCOMES:
Change from Baseline in Coping Strategies Measured by the Brief COPE at Week 10 | From baseline (Week 0) to Week 10 (end of intervention)
  The Brief Coping Orientation to Problems Experienced Inventory (Brief COPE) is a 28-item self-report questionnaire used to assess a person's coping strategies in response to stress. The Brief COPE includes 14 subscales, each with 2 items, scored on a 4-point Likert scale with scores ranging from 0 to 3. Whether higher scores are better or worse depends on the subscale being interpreted.
Change from Baseline in Religious Coping Strategies Measured by the Brief RCOPE at Week 10 | From baseline (Week 0) to Week 10
  The Brief Religious Coping Scale (Brief RCOPE) is designed to assess the extent to which individuals use religious coping in response to stress. The 14 items measure both positive and negative forms of religious coping. Items are on a 4-point Likert scale that ranges from 1 to 4. Higher PRC scores indicate greater use of positive religious coping. Higher NRC scores indicate greater use of negative religious coping.
Change from Baseline in Depression Symptoms Measured by the PHQ-8 at Week 10 | From baseline (Week 0) to Week 10
  The Patient Health Questionnaire-8 (PHQ-8) is an 8-item self-report measure of depression symptoms. Items are on a 4-point Likert scale that ranges from 0 to 3. Total scores range from 0 to 24. Higher scores indicate worse outcomes, i.e., more severe depressive symptoms.
Change from Baseline in Perceived Social Support Measured by the MSPSS at Week 10 | From baseline (Week 0) to Week 10
  The Multidimensional Scale of Perceived Social Support (MSPSS) measures improvement in perceived support from family, friends, and community. 12 items total, each rated on a 7-point Likert scale from 1 to 7. Higher scores indicate greater perceived social support.
Change from Baseline in Posttraumatic Growth Measured by the PTGI at Week 10 | From baseline (Week 0) to Week 10
  The Posttraumatic Growth Inventory (PTGI) assesses positive psychological changes experienced as a result of struggling with highly challenging life circumstances or trauma. 21 items. Each item is scored using a 6-point Likert scale ranging from 0 to 5. Higher scores indicate greater perceived posttraumatic growth.
Change from Baseline in Perceived Social Support Measured by the SCSSS at Week 10 | From baseline (Week 0) to Week 10
  The Spiritual Connectedness Subscale of the Spirituality Scale (SCSSS) assesses a person's perceived connection with the sacred, divine, or transcendent. 5 items total, each rated on a 5-point Likert scale from 1 to 5. Higher scores reflect greater spiritual connectedness.

OTHER OUTCOMES:
Change from Baseline in Group Cohesion Measured by the Group Climate Questionnaire (Sista Circle Edition) at Week 10 | From baseline (Week 0) to Week 10
  Group Climate Questionnaire (Sista Circle Edition) - Adapted from the GCQ (MacKenzie, 1983). Evaluates participants' perceptions of group engagement, conflict, and avoidance within the Sista Circle support groups. 10 items, each rated on a 5-point Likert scale, ranging from 1 to 5. Higher scores in Engagement suggest a constructive group climate, while higher scores in Conflict and Avoidance may indicate challenges within the group dynamics
Change from Baseline in Afrocultural Communal Orientation Measured by the Revised Communalism Scale at Week 10 | From baseline (Week 0) to Week 10
  The Revised Communalism Scale is a psychometric tool used to assess the degree to which individuals endorse communal values, such as interdependence, collective responsibility, and social connectedness, particularly within African American cultural contexts. 5-point Likert scale ranging from 1 to 5.
  Higher scores indicate stronger endorsement of communal values.
Change from Baseline in Whole Person Health Measured by the Whole Person Health Index (WPHI) at Week 10 | From baseline (Week 0) to Week 10
  The WPHI is a multidimensional assessment tool designed to evaluate whole-person health, recognizing the interconnectedness of mind, body, spirit, and community. Nine Items are rated on a Likert-type scale, ranging from 1 to 5. Higher scores indicate greater well-being or more consistent engagement in health-promoting behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Serenity Haven, Lithonia, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared due to the sensitive nature of grief-related experiences and the small sample size, which increases the risk of deductive disclosure even after de-identification. The study population-middle-aged Black women who have experienced the loss of a close loved one-represents a highly specific and vulnerable group. To protect participant confidentiality and respect the culturally sensitive context of the study, data sharing is not planned.

REFERENCES:
- [Background] Jones, M. K., Davis, S. M., & Gaskin-Cole, G. (2023). An integrative review of sistah circles in empirical research. Psychology of Women Quarterly, 47(2), 159-179.
- [Background] Neal-Barnett A, Stadulis R, Murray M, Payne MR, Thomas A, Salley BB. Sister Circles as a Culturally Relevant Intervention for Anxious African American Women. Clin Psychol (New York). 2011 Sep;18(3):266-273. doi: 10.1111/j.1468-2850.2011.01258.x. PMID 22081747
- [Background] Jones, M. K., Gaskin-Cole, G., & Reynolds, A. (2023). Masks off: A community-based psychoeducational group intervention with Black women. The Journal for Specialists in Group Work, 48(3), 212-228.
- [Background] DiGuiseppi G, Rodriguez A, Qureshi N, Zeng C, Coulter ID, Hays RD, Herman PM, Edelen MO. Measuring Whole Person Health: A Scoping Review. J Integr Complement Med. 2025 Aug;31(8):684-704. doi: 10.1089/jicm.2024.0817. Epub 2025 Apr 3. PMID 40180567
- [Background] Brown M, Glendenning A, Hoon AE, John A. Effectiveness of Web-Delivered Acceptance and Commitment Therapy in Relation to Mental Health and Well-Being: A Systematic Review and Meta-Analysis. J Med Internet Res. 2016 Aug 24;18(8):e221. doi: 10.2196/jmir.6200. PMID 27558740
- [Background] Arnold KT, Mandell DS, Hankerson SH. Implementing a Grief Support Program in a Black Church to Support the Mental Health Needs of People in Bereavement. Psychiatr Serv. 2025 Jan 1;76(1):105. doi: 10.1176/appi.ps.20240259. Epub 2024 Oct 23. No abstract available. PMID 39439280